CLINICAL TRIAL: NCT07381244
Title: Validity, Reliability, and Clinical Correlates of Immersive Virtual Reality Adaptation of the Five Times Sit-to-stand Test and Timed up and go Tests in Women With Fibromyalgia Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Zehra KORKUT, Principal Investigator, Selcuk University
Other Study IDs: ZKORKUT_fibromiyalji
Record Dates: First submitted 2026-01-16; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia Syndrome
Keywords: Validity, reliability; fibromyalgia syndrome; virtual reality
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fibromyalgia syndrome (FMS) is a chronic rheumatic condition characterized by widespread pain, fatigue, and functional impairments that negatively affect physical activity levels, muscle strength, balance, and functional mobility. These impairments may lead to reduced functional capacity and increased sedentary behavior. Therefore, objective assessment of mobility, balance, and functional performance is essential in individuals with FMS.

Performance-based tests such as the Five Times Sit-to-Stand Test (5xSTS) and the Timed Up and Go (TUG) test are commonly used to evaluate lower extremity muscle function, balance, and functional mobility due to their simplicity, feasibility, and clinical relevance. Recently, virtual reality (VR)-based assessment methods have emerged as a standardized and objective approach for evaluating functional performance.

This study aims to investigate the feasibility and measurement properties of virtual reality-based adaptations of the 5xSTS and TUG tests in individuals with fibromyalgia syndrome using a head-mounted VR system. Findings from this study are expected to contribute to the clinical use of VR technology in mobility and balance assessment in individuals with FMS.

ELIGIBILITY:
Inclusion Criteria:

* • Having been diagnosed with FMS according to the American Rheumatology Association (ARB) 1990 classification criteria,

  * Being female between the ages of 30-60
  * Having the cognitive ability to understand the instructions
  * Being a volunteer

Exclusion Criteria:

* • Severe physical disability

  * Rheumatological/neurological diseases
  * Any musculoskeletal problem (fracture, deformity, sprain)
  * Malignancy
  * Severe cognitive impairment
  * Pregnancy

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will include adult individuals diagnosed with fibromyalgia according to established diagnostic criteria. Participants will be recruited from outpatient clinics and through announcements. All participants will be able to walk independently and will voluntarily agree to participate in the study. Demographic and clinical characteristics, physical performance, muscle strength, balance, physical activity level, and pain severity will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Performans evaluation | Baseline and 7 days later (test-retest interval).
  Performance outcomes will be assessed using the Five Times Sit-to-Stand Test (5xSTS) and the Timed Up and Go (TUG) test. These tests are widely used functional performance measures with established validity and reliability.
  In this study, virtual reality (VR) adaptations of both tests will also be applied. Participants will enter the testing environment using a VR headset, and test protocols will be conducted in the same manner as the conventional applications. The VR-based assessments will follow standardized procedures equivalent to the traditional versions of the 5xSTS and TUG tests.

SECONDARY OUTCOMES:
Hand Grip Strength | Baseline
  Hand grip strength will be measured in a seated position following standardized testing posture, with the shoulder adducted and in neutral rotation, the elbow flexed to 90 degrees, the forearm supported in mid-rotation, and the wrist in a neutral position. Measurements will be obtained from the dominant hand using a handheld dynamometer. Participants will be instructed to perform a maximal voluntary contraction. Three trials will be conducted with 15-second rest intervals, and the highest value will be recorded in kilograms (kg).
Knee extension muscle strength | baseline
  Knee extension muscle strength will be measured using a handheld dynamometer in a seated position with the hip and knee flexed to 90 degrees. The lower legs will hang freely, and the arms will be crossed over the chest. The dynamometer will be positioned perpendicular to the leg, 1-2 cm proximal to the malleoli, with stabilization applied at the thigh. Three measurements will be obtained, and the highest value will be recorded in kilograms (kg)
Physical Activity Level | baseline
  Physical activity level will be assessed using the 7-item short form of the International Physical Activity Questionnaire. The questionnaire evaluates time spent sitting, walking, moderate-intensity activities, and vigorous-intensity activities during the previous 7 days. Duration (minutes) and frequency (days) of each activity will be recorded. Total physical activity score will be calculated by multiplying activity duration by the corresponding metabolic equivalent (MET) value and summing all activity scores. Physical activity levels will be classified as physically inactive (<600 MET-min/week), minimally active (600-3000 MET-min/week), or active (>3000 MET-min/week).
Single-Leg Balance Test Time | baseline
  Balance will be assessed using the single-leg balance test under eyes-open and eyes-closed conditions. Participants will stand on the dominant leg with the arms crossed over the chest while the contralateral leg is lifted from the ground with the knee flexed to approximately 45 degrees. Timing will begin once the test position is achieved. The test will be terminated if the arms or the non-stance leg are used for support or when the maximum duration of 30 seconds is reached. Time will be recorded in seconds. Each condition will be repeated three times, and the best performance will be recorded. The same procedure will be applied to the nondominant leg

IPD SHARING:
Plan to Share IPD: No